CLINICAL TRIAL: NCT03243604
Title: Cardiotoxicity of Abiraterone in the National French Pharmacovigilance Database and in the European Clinical Trials Database (EudraCT)
Brief Title: cARdiotoxicity Profile of aBIraTeRone in prostAte Cancer : a pharmacoviGilancE Study
Acronym: ARBITRAGE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-17-08
Record Dates: First submitted 2017-07-20; First posted 2017-08-09 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation and Flutter; Tachycardia, Supraventricular; Cardiac Failure
Keywords: Cardiotoxicity; abiraterone acetate; androgen antagonist
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Tachycardia, Supraventricular; Heart Failure; Cardiotoxicity | interventions — Gonadal Steroid Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: L02 (sex hormones used in treatment of neoplastic diseases) and G03 (sex hormones) — Androgen-deprivation therapies including L02 (sex hormones used in treatment of neoplastic diseases), and G03 (sex hormones)

SUMMARY:
Abiraterone associated with prednisone is used in prostate cancer. Abiraterone is a selective small-molecule inhibiting cytochrome P450 17A1 (CYP17A1), a key enzyme in androgen synthesis.

CYP17A inhibition is also responsible for mineral corticosteroid related adverse events as hypokaliemia, fluid retention, and hypertension. Primary hyperaldosteronism is associated with cardiovascular toxicities such as atrial fibrillation and cardiac failure. Other androgen-deprivation therapies are not associated with increased mineral corticosteroid level.

This study investigates reports of cardiovascular toxicities for treatment including L02 (sex hormones used in treatment of neoplastic diseases), and G03 (sex hormones) used in prostate cancer in the French pharmacovigilance database and in the EudraCT database.

DETAILED DESCRIPTION:
Due to its peculiar pharmacology, abiraterone is potentially associated with more cardiotoxicity as compared to other androgen-deprivation therapies. This study investigates the main characteristics of patients affected by cardiovascular side effects of which supraventricular arrhythmias (including atrial fibrillation, atrial flutter, supraventricular tachycardia), and cardiac failure imputed to drugs classified as L02, and G03 according to anatomical therapeutic chemical (ATC) classification. A causality assessment according to the World Health Organization-The Uppsala Monitoring Centre (WHO-UMC) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the French pharmacovigilance database from 01/01/1985 to 16/05/2017
* Case reported in the EudraCT database to May 2017
* Adverse event reported were including the MedDRA terms: SOC Cardiac Disorders; SOC Vascular Disorders; HLT Death, Sudden Death; HLGT Water, electrolyte and mineral investigations; HLGT Cardiac and vascular investigations (excl enzyme tests); and PT Syncope.
* Patients treated with hormonal therapies included in the ATC L02, and G03

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: The population is selected in the French pharmacovigilance database and EudraCT database from 01/01/1985 to May 2017 and included patients treated with hormonal therapies included in the ATC L02, and G03
Sampling Method: Non-Probability Sample
Enrollment: 1717 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Analysis of disproportionality of reports for cardiotoxicity associated with abiraterone as compared to enzalutamide by performing a case- non-case study | 2 months
  Analysis of disproportionality of reports for cardiotoxicity associated with abiraterone as compared to enzalutamide by performing a case- non-case study

SECONDARY OUTCOMES:
Compare the reporting of suspected drug-induced supraventricular arrhythmias with abiraterone as compared to enzalutamide by performing a disproportionality analysis | 2 months
  Compare the reporting of suspected drug-induced supraventricular arrhythmias with abiraterone as compared to enzalutamide by performing a disproportionality analysis
Compare the reporting of drug-induced cardiac failure with abiraterone as compared to enzalutamide by performing a disproportionality analysis | 2 months
  Compare the reporting of drug-induced cardiac failure with abiraterone as compared to enzalutamide by performing a disproportionality analysis
Compare the reporting of drug-induced cardiac failure and/or supraventricular arrhythmias with abiraterone as compared to other androgen-deprivation therapies by performing a disproportionality analysis | 2 months
  Compare the reporting of drug-induced cardiac failure and/or supraventricular arrhythmias with abiraterone as compared to other androgen-deprivation therapies by performing a disproportionality analysis
Description of other mineralocorticoid related adverse events (hypokaliemia, fluid retention, and hypertension) when the cardio toxicity occurs | 2 months
  Description of other mineralocorticoid related adverse events (hypokaliemia, fluid retention, and hypertension) when the cardio toxicity occurs
Description of the population of patients having a cardio-vascular adverse event | 2 months
  Description of the population of patients having a cardio-vascular adverse event
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | 2 months
  Description of the duration of treatment when the toxicity happens (role of cumulative dose)
Description of the drug-drug interactions associated with adverse events | 2 months
  Description of the drug-drug interactions associated with adverse events
Causality assessment of reported cardiovascular events according to the WHO-UMC system | 2 months
  Causality assessment of reported cardiovascular events according to the WHO-UMC system

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Régional de Pharmaco-vigilance - Paris, Pitié-Salpétrière, Paris, Île-de-France Region, France